CLINICAL TRIAL: NCT05378139
Title: WARD Prospective Study - Continuous Wireless Monitoring of Vital Signs and Automated Alerts in Participants at Home and During Hospitalization
Brief Title: Continuous Wireless Monitoring of Vital Signs and Automated Alerts in Participants at Home and During Hospitalization
Status: Recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Katja Kjær Grønbæk, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: 2203648
Record Dates: First submitted 2022-04-07; First posted 2022-05-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-07

CONDITIONS: Surgical Complication; Pulmonary Disease; Hematologic Diseases; Oncology; Cardiac Disease; Infections
MeSH Terms: conditions — Lung Diseases; Hematologic Diseases; Neoplasms; Heart Diseases; Infections | interventions — Vital Signs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Vital signs measurements with new app — Patients vital signs are monitored through an app for the nurses to use

SUMMARY:
The primary aim of this study is to test and assess the implementation and effectiveness of continuous wireless vital signs monitoring with real-time alerts on:

The frequency of patients monitored with adequate data quality as adequate clinical user satisfaction in the initial versus the last part of the trial (primary outcome).

DETAILED DESCRIPTION:
Over the last years, the applicants and research team partners have developed the WARD (Wireless Assessment of Respiratory and circulatory Distress) project, using continuous wireless monitoring of vital signs and artificial intelligence algorithms for data interpretation in high-risk patient admitted to medical and surgical wards. The WARD project combines continuous measurements of 10 different physiological modalities with machine learning to develop the WARD-Clinical Support System (WARD-CSS), based on multiple intelligent algorithms, that automatically monitors, interprets, predicts and alert clinical staff. Through a mobile device with a purpose-built Graphic User Interface (GUI), the WARD-CSS stimulates human-machine interaction to improve the monitoring of high-risk hospitalized patients.

The WARD project has hitherto proven an unmet need for continuous monitoring and the potential for automatic detection and prediction of physiological deterioration events. Specifically, observational pilot studies of both patients with acute exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD) and postoperative abdominal cancer surgery patients have shown that episodes of desaturation, tachycardia, tachypnea, and bradypnea are much more frequently detected using continuous vital signs monitoring than with existing Early Warning Score (EWS) systems.

Ongoing investigations will determine the efficacy in two very selected populations of high-risk surgical patients and acutely ill medical patients with severe disease. This study will investigate the WARD-systems' implementation, and effectiveness of use and impact in a cohort of patientparticipants admitted

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥18 years)
* Patients assessed by the clinical staff as having an acute condition with risk for clinical deterioration and being either at home (with no apparent need for hospitalization), and/or in hospital OR
* Patients at either at home before, in-hospital and/or after hospitalization for elective major surgery, defined as surgery lasting more than one hour under general- or regional anaesthesia

Exclusion Criteria:

* The participant expected not to cooperate with study procedures.
* Allergy to plaster or silicone.
* Having pacemaker or Implantable Cardioverter Defibrillator (ICD) device.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assessed by the clinical staff as having an acute condition with risk for clinical deterioration and being either at home (with no apparent need for hospitalization), and/or in hospital
  OR
  Patients at either at home before, in-hospital and/or after hospitalization for elective major surgery, defined as surgery lasting more than one hour under general- or regional anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 3095 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Data quality | 30 days
  The number (frequency) of patients having adequate data quality (defined as at least 60% of the monitoring time with simultaneous recording of SpO2, respiratory rate, heart rate)
user satisfaction | 30 days
  Number of users with adequate clinical user satisfaction (defined as the nurse in charge of the patient at the end of monitoring answers "Agree" or "Strongly agree" to the question "WARD-monitoring was beneficial for monitoring of vital signs in this patientparticipant (response options: Strongly Disagree - Disagree - Neutral - Agree - Strongly Agree)).

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided upon reasonable request